CLINICAL TRIAL: NCT03741387
Title: Saving a Life or Preventing a Death: the Effect of Message Framing on Blood Donation Among Rh Negative Donors
Brief Title: The Effect of Message Framing on Blood Donation-Study 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Blood Center (Other Government)
Responsible Party: Principal Investigator, OUYANG Jian, MS, Guangzhou Blood Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Message Framing effect 2
Record Dates: First submitted 2018-11-11; First posted 2018-11-14 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Rh Negative Blood Donor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gain-frame questionnaire (Experimental): Questionnaire included a picture of a patient lying in bed entitled "Will you save his life?" Donors in this group will answer the questions about attitude of saving patients' lives.
  Interventions: Other: Gain-frame questionnaire
- Loss-frame questionnaire (Experimental): Questionnaire included a picture of a patient lying in bed entitled "Will you prevent him from death?" Donors in this group will answer the questions about the attitude of preventing patients from death.
  Interventions: Other: Loss-frame questionnaire

INTERVENTIONS:
Other: Gain-frame questionnaire — Questionnaires focusing on the attitude of saving patients' lives were given to Rh negative blood donors in this group.
  Arms: Gain-frame questionnaire
Other: Loss-frame questionnaire — Questionnaires focusing on the attitude of preventing patients from death were given to Rh negative blood donors in this group.
  Arms: Loss-frame questionnaire

SUMMARY:
Rh negative blood group is a rare blood group in China, as it only accounts for 0.3-0.4 percent of the Han population. Therefore, low inventory is often found in blood collection and supply agencies in many regions in China. In order to assess the effects of the gain-versus-loss framing message on blood donation among Rh negative donors, we designed two kinds of self-administered, standardized and structured questionnaires. In addition of the basic socio-demographic characteristics, one questionnaire includes the questions which survey the attitude of saving patients lives, and the other was to survey the attitude of preventing patients from death. The questionnaires were randomly sent to Rh negative blood donors.

ELIGIBILITY:
Inclusion Criteria:

* Rh negative blood donors who have donated blood between 2016 and 2018.

Exclusion Criteria:

* People who are Rh negative blood type but never have donated blood.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 795 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2019-03-21 (Actual); Study Completion 2019-03-21 (Actual)

PRIMARY OUTCOMES:
The differences of attitude towards different massage framing | 1 day
  After participants view the picture in their questionnaires, they would answer the questions about attitude of saving patients' lives or preventing patients from death.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Blood Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No